CLINICAL TRIAL: NCT06166212
Title: Changes in Angle Kappa and Corneal Back Elevations After Laser in Situ Keratomileusis in Myopic Astigmatism
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohamed Elsaiid, Ophthalmology Specialist, Ain Shams University
Other Study IDs: angle K relation e astigmatism
Record Dates: First submitted 2023-11-19; First posted 2023-12-12 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Refractive Errors
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases with high myopic astigmatism: Cases having myopic astigmatism more than 1.5 diopter
- Cases with not high astigmatism: Cases having astigmatism less than 1.5 diopter

SUMMARY:
Refractive errors and corneal astigmatism are associated with changes in angle kappa and corneal back elevation at the thinnest point in Pentacam.

The purpose of this study is to track:

The effect of anterior corneal astigmatism treatment on angle kappa and corneal back elevation.

DETAILED DESCRIPTION:
This prospective observational study will be settled in Ain Shams University Hospital, Cairo, Egypt.

ELIGIBILITY:
Inclusion Criteria:

Myopic astigmatism

Exclusion Criteria:

Corneal scar

Ages: 18 Years to 40 Years | Sex: All
Age Groups: Adult
Study Population: 2 groups
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Track changes in angle kappa | through study completion, an average of 2 years
  Track changes in angle kappa with changes in corneal astigmatism

DOCUMENTS (1):
  • Study Protocol (2023-12-03): https://cdn.clinicaltrials.gov/large-docs/12/NCT06166212/Prot_000.pdf